CLINICAL TRIAL: NCT00804271
Title: Open Label, Single-Arm, Multi-Centre, Study to Validate a New Alzheimer's Disease Scale in Patients With DAT, Treated With Memantine
Brief Title: Memantine and Validation of a New Alzheimer's Disease Scale
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MRZ 90001/AD/3001; EudraCT No. 2008-005144-16
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Other)
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — memantine tablets, OD, 12 weeks
  Other Names: Axura

SUMMARY:
To validate a new Alzheimer's Disease scale against other rating tools in subjects with dementia of Alzheimer's type, treated with memantine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease consistent with NINCDS-ADRDA criteria or with DSM IV TR criteria for Dementia of Alzheimer's type.
* Signed informed consent prior to the initiation of any study specific procedures.
* Sight and hearing (a hearing aid is permitted) are sufficiently good to allow the undertaking of study-related procedures and psychometric tests.

Exclusion Criteria:

* Evidence of clinically significant and active pulmonary, gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease.
* Intake of any medication that is contra-indicated in combination with memantine.
* History of severe drug allergy, or hypersensitivity, or patients with known hypersensitivity to ingredients of memantine or lactose.
* Known or suspected history of alcoholism or drug abuse within the past 2 years.
* Current or previous treatment with memantine or participation in an investigational study with memantine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Validation of new scale regarding content, reliability and responsiveness for DAT symptoms | at post baseline visit

SECONDARY OUTCOMES:
Assessment of treatment response and correlation of new scale against ADAScog, SIB, NPI, DAD. | at a post baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Vjera Holthoff, MD, Principal Investigator — University Clinic Gustav Carus Dresden, Germany
Locations (1):
- University Clinic Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Result] Holthoff V, Ferris S, Gauthier S, Ihl R, Robert P, Winblad B, Sternberg K, Tennigkeit F; ROSA Study Group. Memantine effects measured with the Relevant Outcome Scale for Alzheimer's disease in an open-label, single-arm, multicenter clinical study. Int J Geriatr Psychiatry. 2013 Feb;28(2):164-72. doi: 10.1002/gps.3805. Epub 2012 Apr 11. PMID 22492589
- [Result] Holthoff VA, Ferris S, Ihl R, Robert P, Winblad B, Gauthier S, Sternberg K, Tennigkeit F. Validation of the relevant outcome scale for Alzheimer's disease: a novel multidomain assessment for daily medical practice. Alzheimers Res Ther. 2011 Jul 6;3(5):27. doi: 10.1186/alzrt89. PMID 21914212